CLINICAL TRIAL: NCT06701110
Title: Pharmacokinetics and Mass Balance Study of WX-081 (Sudapyridine) in Healthy Chinese Volunteers
Brief Title: Pharmacokinetic Study of Sudapyridine（WX-081）in Healthy Chinese Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JYP0081M102
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: TB
MeSH Terms: interventions — sudapyridine

STUDY DESIGN:
Intervention Model Description: This study involves a single cohort of healthy male volunteers receiving a single oral dose of [U-14C] WX-081 to evaluate pharmacokinetics, metabolism, and mass balance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Oral Dose of [U-14C] WX-081 (Experimental): Participants will receive a single oral dose of approximately 450 mg (100 μCi) of [U-14C] WX-081. The study involves collecting biological samples, including blood, plasma, urine, and feces, at specified time points to evaluate pharmacokinetics, metabolism, mass balance, and excretion pathways.
  Interventions: Drug: [U-14C] WX-081

INTERVENTIONS:
Drug: [U-14C] WX-081 — A single oral dose of approximately 450 mg (100 μCi) of [U-14C] WX-081 will be administered to healthy male volunteers. The study will involve pharmacokinetic assessments, including metabolism, mass balance, and excretion pathways, through the collection of biological samples such as blood, plasma, urine, and feces.
  Other Names: Sudapyridine

SUMMARY:
This single-center, open-label, non-randomized study aims to evaluate the pharmacokinetics, mass balance, and metabolic pathways of WX-081 (Sudapyridine) following a single oral dose of [U-14C] WX-081 in healthy Chinese male volunteers. A total of 6-10 subjects will be enrolled to obtain complete samples and data from at least six participants. Biological samples, including blood, plasma, urine, and feces, will be collected over a specified time period. The study will assess pharmacokinetic parameters, excretion pathways, and identify major metabolites contributing to over 10% of plasma exposure.

DETAILED DESCRIPTION:
The study involves healthy male volunteers who will receive a single oral dose of [U-14C] WX-081 containing approximately 450 mg (100 μCi) after fasting overnight. Samples of blood, plasma, urine, and feces will be collected during an intensive phase (up to 504 hours post-dose) and a sparse phase (up to 51 days). Pharmacokinetic and excretion parameters will be calculated, and metabolic pathways will be determined via radiolabeled metabolite profiling. Volunteers will follow pre-specified dietary and procedural requirements, including pre-dose baseline assessments and post-dose fasting. Adjustments to sample collection duration or early termination will be made based on phase-specific results. Safety monitoring will continue until sample collection is complete.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males. Age: 18-45 years (inclusive). Body weight: BMI between 19.0 and 26.0 kg/m² (inclusive), with body weight not less than 50.0 kg.

Voluntarily signed the informed consent form. Able to communicate effectively with investigators and comply with the study protocol.

Exclusion Criteria:

* Clinically significant abnormalities identified through physical examination, vital signs, laboratory tests (e.g., blood count, biochemistry, troponin, coagulation function, urinalysis, fecal occult blood), thyroid function, 12-lead ECG, chest X-ray, rectal examination, or abdominal ultrasound (liver, gallbladder, pancreas, spleen, kidney).

Prolonged corrected QT interval (QTcF) > 450 msec on 12-lead ECG. Positive results for hepatitis B surface antigen (HBsAg or HBeAg), hepatitis C antibody (HCV-Ab), syphilis antibody, or HIV antigen/antibody (HIV-Ag/Ab).

Use of drugs that inhibit or induce hepatic enzymes or transporters within 30 days prior to screening.

Use of prescription or over-the-counter medications, herbal remedies, or dietary supplements (e.g., vitamins, calcium) within 14 days prior to screening.

Any clinically significant disease or condition that may affect study results, including but not limited to cardiovascular, respiratory, endocrine, neurological, gastrointestinal, urinary, hematological, immune, psychiatric, or metabolic disorders.

Conditions that could affect drug absorption, such as a history of gastric surgery (e.g., gastrectomy, gastric bypass), gallbladder removal, or inflammatory bowel disease.

History of organic heart disease, heart failure, myocardial infarction, angina, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, long QT syndrome, or family history of sudden cardiac death due to cardiac reasons.

Major surgery within 6 months prior to screening or incomplete surgical wound healing.

Known hypersensitivity or allergy to two or more substances, or potential allergy to the investigational drug or its excipients (e.g., lactose, low-substituted hydroxypropyl cellulose, sodium lauryl sulfate, silicon dioxide, magnesium stearate).

Hemorrhoids or perianal conditions with regular or current rectal bleeding.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative Excretion Rate of Total Radioactivity in Urine | Up to Day 51 post-dose.
  The cumulative percentage of total radioactivity excreted in urine and feces after a single oral dose of [U-14C] WX-081 in healthy male volunteers.
Cumulative Excretion Rate of Total Radioactivity in Feces | Up to Day 51 post-dose.
  The cumulative percentage of total radioactivity excreted in feces after a single oral dose of [U-14C] WX-081 in healthy male volunteers.

SECONDARY OUTCOMES:
Identification and Percentage of Major Metabolites in Plasma, Urine, and Feces | Up to Day 51 post-dose
  The percentage of total radioactivity in plasma attributable to the parent drug and its metabolites (≥10% of total AUC) and the percentage of dose excreted in urine and feces as the parent drug and metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China